CLINICAL TRIAL: NCT00478283
Title: Perspectives and Attitudes on the Use of Adjuvant Chemotherapy and Hormonal Therapy in Older and/or Frail Women: A Survey of Oncologists and Geriatricians
Brief Title: Views and Attitudes of Oncologists and Geriatricians on the Use of Chemotherapy and Hormone Therapy in Treating Older and/or Frail Women With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Arti Hurria MD, City of Hope Medical Center
Purpose: Health Services Research
Other Study IDs: CDR0000540280; P30CA033572 (NIH); CHNMC-06187
Record Dates: First submitted 2007-05-23; First posted 2007-05-24 (Estimated); Last update posted 2010-02-09 (Estimated); Status verified 2010-02

CONDITIONS: Breast Cancer
Keywords: breast cancer
MeSH Terms: conditions — Breast Neoplasms

INTERVENTIONS:
Other: survey administration

SUMMARY:
RATIONALE: A patient's age, health, and ability to perform daily activities may affect which treatment options are offered by doctors to older and/or frail women with breast cancer.

PURPOSE: This clinical trial is studying the views and attitudes of oncologists and geriatricians on the use of chemotherapy and hormone therapy in treating older and/or frail women with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the attitudes and perspectives of 150 oncologists and 150 geriatricians or primary care providers regarding the adjuvant treatment of older women with breast cancer of varying ages, health, and functional status.
* Determine whether homogeneity exists in treatment recommendations.
* Determine the relative impact of chronological age, baseline health, and functional status on treatment recommendations.

OUTLINE: Participants complete a 25-minute online survey regarding their treatment recommendations for older women with breast cancer of varying ages, health, and functional status.

PROJECTED ACCRUAL: A total of 300 participants will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Participants must meet 1 of the following criteria:

  * Oncologist:

    * Must have been in practice ≥ 2 years
    * Must have ≥ 25 postmenopausal breast cancer patients on adjuvant hormonal therapy
    * Cannot work for an advertising agency, market research company, manufacturer or distributor of pharmaceutical products, a pharmacy, drug store, or the FDA
  * Geriatrician:

    * Must have been in practice ≥ 2 years
    * Must be a general practitioner, family practitioner, internal medicine specialist, or geriatrician and received a certificate of added qualification in geriatric medicine and/or treating at least 5 postmenopausal patients who have a history of breast cancer or are currently undergoing treatment for breast cancer
    * Cannot work for an advertising agency, market research company, manufacturer or distributor of pharmaceutical products, a pharmacy, drug store, or the FDA

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2006-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Attitudes and perspectives of health professionals
Homogeneity of treatment recommendations
Relative impact of chronological age, baseline health, and functional status on treatment recommendations

CONTACTS AND LOCATIONS:
Overall Officials: Arti Hurria, MD, Principal Investigator — City of Hope Comprehensive Cancer Center